CLINICAL TRIAL: NCT02705196
Title: Phase I/IIa Trial Evaluating Safety of LOAd703, an Armed Oncolytic Adenovirus for Pancreatic Cancer
Brief Title: LOAd703 Oncolytic Virus Therapy for Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lokon Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LOKON001
Record Dates: First submitted 2016-02-15; First posted 2016-03-10 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer
Keywords: oncolytic; adenovirus; pancreatic; cancer; LOKON; LOAd703
MeSH Terms: conditions — Pancreatic Neoplasms; Adenoviridae Infections; Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 Intratumoral LOAd703 (Experimental): Patients will receive gemcitabine intravenously at a dose of 1000mg/m2 + nab-paclitaxel 125 mg/m2 as per hospital standards. One cycle will be one dose of gemcitabine +nab-paclitaxel given on days 1, 8, and 15 of a 28 day cycle. LOAd703 will be given every other week for 6 doses starting on day 15 of the first cycle of chemotherapy. There is an option for an additional 6 doses if patients benefit from treatment.
  The following LOAd703 doses will be evaluated:
  Dose level 1: 5 X 10^10 viral particles per treatment Dose level 2: 1 X 10^11 viral particles per treatment Dose level 3: 5 X 10^11 viral particles per treatment
  Interventions: Genetic: delolimogene mupadenorepvec; Drug: gemcitabine; Drug: nab-paclitaxel
- Arm 2: Intratumoral LOAd703 + atezolizumab (Experimental): Patients will receive gemcitabine intravenously at a dose of 1000mg/m2 + nab-paclitaxel 125 mg/m2 as per hospital standards. One cycle will be one dose of gemcitabine +nab-paclitaxel given on days 1, 8, and 15 of a 28 day cycle. LOAd703 will be given every other week for 6 doses starting on day 15 of the first cycle of chemotherapy. There is an option for an additional 6 doses if patients benefit from treatment. A fixed dose of atezolizumab 1680 mg will be given every 4 weeks on day 1 of each chemotherapy cycle.
  Patients will be assigned to the following LOAd703 doses:
  Dose level 1: 1 X 10^11 viral particles per treatment Dose level 2: 5 X 10^11 viral particles per treatment
  Interventions: Genetic: delolimogene mupadenorepvec; Drug: gemcitabine; Drug: nab-paclitaxel; Biological: atezolizumab

INTERVENTIONS:
Genetic: delolimogene mupadenorepvec — oncolytic virus encoding TMZ-CD40L and 4-1BBL
  Other Names: LOAd703
Drug: gemcitabine — chemotherapy
  Other Names: Gemzar
Drug: nab-paclitaxel — chemotherapy
  Other Names: Abraxane
Biological: atezolizumab — anti-PD-L1 antibody
  Other Names: Tecentriq
  Arms: Arm 2: Intratumoral LOAd703 + atezolizumab

SUMMARY:
The purpose of this study is to see if LOAd703 (an oncolytic adenovirus) can be safely given to patients with pancreatic cancer. The study will also evaluate whether or not intratumoral injection of LOAd703 will support current standard of care treatment to reduce the size of the tumor and improve survival of the patients.

Adenoviruses are known as the "common cold" virus and most individuals have had multiple infections during their lifetime. Oncolytic adenoviruses are adenoviruses that are modified so they cannot multiply and spread (known as replicating) properly in normal (e.g. healthy) cells, but instead, they infect and replicate very well in cancer cells. This strong replication leads to the death of the cancer cell. Oncolytic viruses have been evaluated in multiple clinical trials for cancer treatment during the past decade and been proven safe. It is common to have a fever the first day or two after virus injection since the immune system will react to the virus infection. The immune system can also kill cancer cells but to do so it needs to be properly stimulated. Oncolytic viruses alone do not seem to be strong enough to activate clinically relevant anti-cancer responses. However, it is thought that if additional immune system stimulators are added to the oncolytic viruses they may be able to result in clinical relevant antic-cancer responses.

LOAd703 is an oncolytic adenovirus that has been modified to include additional immune system stimulators. Specifically, genes that stimulate the immune system have been added to the oncolytic adenovirus. Once the oncolytic adenovirus infects the cancer cells, the genes will be expressed, resulting in activation of the immune response so it can attack and kill cancer cells.

In this study, LOAd703 will be given by intratumoral injections. It will be given in addition to standard of care treatment with gemcitabine and nab-paclitaxel +/- the anti-PD-L1 antibody atezolizumab. Because this is an experimental therapy, there will be extra visits for disease monitoring and samples accordingly to the detailed information below. The LOAd703 is an investigational agent not approved by the FDA.

DETAILED DESCRIPTION:
The research will be conducted at Baylor College of Medicine (BCM) and Baylor St. Luke's Medical Center (BSLMC).

All patients will receive standard of care treatment for their pancreatic cancer. Standard of care treatment will be gemcitabine in combination with nab-paclitaxel given on days 1, 8, and 15 of a 28 day cycle.

Arm 1: LOAd703 treatment will be initiated at day 15 of the first cycle and given every other week for 6 doses. Depending on the location of the tumor the injection of LOAd703 can be given in different ways. The most common route of injection is ultrasound-guided percutaneous injection, but endoscopic ultrasound-guidance will be used for some patients as appropriate. All patients will receive anti-anxiety drugs or sedation as needed for comfort during the procedure. This study evaluates different doses of LOAd703. All patients will receive six injections of LOAd703. If patients in either phase of the study are judged by the investigator to be deriving clinical benefit from LOAd703 once all scheduled injections have been administered, they will be eligible to receive up to 6 additional biweekly doses of LOAd703.

Arm 2: the same procedures as arm 1 in regard to LOAd703. In addition, the arm 2 patients will receive atezolizumab at a fixed dose, every chemotherapy cycle day 1. The treatments can continue until the final follow-up visit.

Follow-up visits: Besides visits to receive treatments, patients will continue to visit BCM/BSLMC or their local doctor for evaluation of health status and side effects. At some visits blood samples will be obtained. Some of the blood samples being obtained are considered standard of care to ensure patient safety for standard of care treatment and the LOAd703 injection. However, some blood and biopsy samples (in applicable patients) will be collected to be analyzed for the presence of LOAd703, atezolizumab tumor markers and immunology markers. The extra blood will be 5-15 ml (3 teaspoonfuls) of blood collected at the screening visit and at eight different time points both during treatment and after treatments are completed. Imaging of the tumor to determine tumor size will be done every two to three months, which is routine for the monitoring of patients with pancreatic cancer. Patients will actively participate in the study for about 9 months when the final follow-up visit will be scheduled (or 12 months if additional doses of LOAD703 are given). After their active participation is completed patients will continue to receive routine care and will be contacted by the study team every 3 months to provide follow up on the status of their disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ductal adenocarcinoma of the pancreas (PDAC).
2. Low tumor burden with at least one lesion that is suitable for image-guided intratumoral injection and needle biopsy.
3. The patient is not eligible for a complete surgical resection of their disease as evaluated by a radiologist and/or surgeon.
4. Patients who may receive the injections endoscopically should be eligible for sedation.
5. The patient must be eligible for standard of care treatment with gemcitabine +nab-paclitaxel.
6. Age ≥ 18 yrs of age
7. Females of childbearing potential must have a negative pregnancy test and agree to use contraception during on-study protocol treatment.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
9. Absolute neutrophil count (ANC) ≥1.0 x 10^9/l, hemoglobin ≥9 g/dl, platelet count ≥ 100 x 10^9/l, prothrombin (INR) <1.5.
10. Adequate hepatic function, with bilirubin < 1.5 x the ULN, and AST and ALT < 2.5 x ULN
11. Adequate renal function with serum creatinine <2 x the ULN or creatinine clearance >30 mL/min
12. The patient must provide informed consent.

Exclusion Criteria:

1. Any concurrent treatment that would compromise the study including but not limited to continuous high dose corticosteroids (>10 mg/day of prednisone equivalence), lymphodepleting antibodies or cytotoxic agents.
2. Treatment with high dose immune inhibitors including lymphotoxic monoclonal antibodies such as alemtuzumab (Campath), or rapamycin/rapalogs or cytotoxic agents within 21 days of registration
3. Treatment with biologic therapy within 21 days of registration.
4. Use of any investigational agents within 21 days of registration.
5. The use of systemic immunostimulatory agents (including, but not limited to, interferons and IL-2) are prohibited within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment and during study treatment because these agents could potentially increase the risk for autoimmune conditions when given in combination with atezolizumab
6. Pregnant or breastfeeding females.
7. Known active hepatitis B or C infection, HIV infection or tuberculosis.
8. Patients with active autoimmune disease or immune deficiency or previous Guillain-Barre syndrome. Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only (e.g. patients with psoriatic arthritis are excluded) are eligible for the study provide all of the following conditions are met:

   * Rash must cover <10% of body surface area
   * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
   * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors or high-potency or oral corticosteroids within the previous 12 months
9. Uncontrolled intercurrent illness including but not limited to psychiatric illness/social situations that in the opinion of the Investigator would compromise compliance of study requirements or put the patient at unacceptable risk.
10. Other malignancies within the past 2 years (not including basal cell carcinoma of the skin, prostate cancer or in situ cervix carcinoma).
11. Moderate to large volume ascites.
12. History of leptomeningeal disease.
13. Uncontrolled pleural effusion, pericardial effusion or ascites requiring recurrent drainage procedures (once monthly or more frequently)
14. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis or evidence of active pneumonitis on screening chest computed tomography (CT) scan. However, history of radiation pneumonitis in the radiation field (fibrosis) is permitted.
15. Unstable angina, uncontrolled cardiac arrhythmia, recent (within 3 months) history of myocardial infarction or stroke or New York Class III/IV congestive heart failure
16. Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment or anticipation of need for a major surgical procedure during the study.
17. Prior allogeneic stem cell or solid organ transplantation.
18. History of severe allergic anaphylactic reactions to chimeric human or humanized antibodies or fusion proteins.
19. Known hypersensitivity to CHO cell products or any component of the atezolizumab formulation.
20. Live attenuated vaccines (e.g. FluMist) are prohibited within 4 weeks prior to initiation of study treatment, during atezolizumab treatment, and for 5 months after the final dose of atezolizumab.
21. Adenovirus-based vaccines (e.g Vaxzevria, known as COVID-19 vaccine Astra Zeneca, J&J Covid-19 vaccine) are prohibited 3 months prior to initation of study treatment, during treatment and 6 months after the final dose of LOAd703

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patient with dose-limiting toxicities (DLTs) as evaluated accordingly to CTCAE 4.0 | 9 months
  Maximum tolerated dose of multiple (6x) image-guided intratumoral injections of LOAd703 at three dose levels in combination with standard of care therapy

SECONDARY OUTCOMES:
Overall Response Rate | 9 months
  To determine the percentage of subjects achieving a partial response or better (according to RECIST 1.1) to repeat doses of LOAd703 (at the highest dose as determined in Phase I) combined with standard of care treatment with and without atezolizumab in pancreatic cancer.
Overall Survival | 6 months post last patient, last visit
  To determine the survival days post study initiation

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Loskog, PhD, Study Chair — Lokon Pharma AB
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Baylor St Luke's Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Musher BL, Rowinsky EK, Smaglo BG, Abidi W, Othman M, Patel K, Jawaid S, Jing J, Brisco A, Leen AM, Wu M, Sandin LC, Wenthe J, Eriksson E, Ullenhag GJ, Grilley B, Leja-Jarblad J, Hilsenbeck SG, Brenner MK, Loskog ASI. LOAd703, an oncolytic virus-based immunostimulatory gene therapy, combined with chemotherapy for unresectable or metastatic pancreatic cancer (LOKON001): results from arm 1 of a non-randomised, single-centre, phase 1/2 study. Lancet Oncol. 2024 Apr;25(4):488-500. doi: 10.1016/S1470-2045(24)00079-2. PMID 38547893
- See also: Sponsors website — http://www.lokonpharma.com